CLINICAL TRIAL: NCT01637454
Title: NORADRENALINE VERSUS TERLIPRESSIN IN THE TREATMENT OF TYPE 2 HEPATORENAL SYNDROME:A RANDOMIZED STUDY
Brief Title: TYPE 2 HEPATORENAL SYNDROME
Acronym: Type2 HRS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Arun Sharma, Clinical Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGIMERIndia
Record Dates: First submitted 2012-06-28; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Safety and Efficacy of Terlipressin and Noradrenaline and Predictive Factors of Response in Type 2 HRS
Keywords: noradrenaline terlipressin type 2 HRS
MeSH Terms: interventions — Norepinephrine; Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terlipressin and Type-2 HRS (Active Comparator): Patients in group A received terlipressin as an intravenous bolus of 0.5 mg every 6 h. If a significant reduction in serum creatinine level (≥1 mg/dL) was not observed during 3-day period, the dose of terlipressin was increased in a stepwise fashion every 3 days to a maximum of 2 mg every 6 hour.
  Interventions: Drug: Noradrenaline; Drug: Terlipressin
- Noradrenaline and Type-2 HRS (Active Comparator): Patients in group B received a continuous infusion of noradrenaline at an initial dose of 0.5 mg/hour, designed to achieve an increase in mean arterial pressure (MAP) of at least 10mmHg or an increase in 4-h urine output to more than 200 mL. When one of these goals was not achieved, the noradrenaline dose increased every 4 hour in steps of 0.5 mg/hour, up to the maximum dose of 3 mg/hour
  Interventions: Drug: Noradrenaline; Drug: Terlipressin

INTERVENTIONS:
Drug: Noradrenaline — Patients in group B received a continuous infusion of noradrenaline at an initial dose of 0.5 mg/hour, designed to achieve an increase in mean arterial pressure (MAP) of at least 10mmHg or an increase in 4-h urine output to more than 200 mL. When one of these goals was not achieved, the noradrenaline dose increased every 4 hour in steps of 0.5 mg/hour, up to the maximum dose of 3 mg/hour
Drug: Terlipressin — Patients in group A received terlipressin as an intravenous bolus of 0.5 mg every 6 h. If a significant reduction in serum creatinine level (≥1 mg/dL) was not observed during 3-day period, the dose of terlipressin was increased in a stepwise fashion every 3 days to a maximum of 2 mg every 6 hour

SUMMARY:
Various vasoconstrictors have shown promising results in the management of type 1 hepatorenal syndrome (HRS). However, there are very few studies on vasopressors in the management of type 2 HRS. Terlipressin has been used commonly; however it is costly and not available in some countries. In the present study, the investigators evaluated safety and efficacy of terlipressin and noradrenaline in the treatment of type 2 HRS

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis with ascites with serum creatinine more than 1.5 mg/dl and less than 2.5 mg/dl
2. Absence of shock, fluid losses and treatment with nephrotoxic drug
3. No improvement in renal function following diuretic withdrawal and plasma volume expansion
4. No ultrasound evidence of renal parenchymal disease or obstructive uropathy 5.Absence of proteinuria more than 500 mg/24 hour

Exclusion Criteria:

1. Patients with history of coronary artery disease
2. Cardiomyopathy
3. Ventricular arrhythmia
4. Obstructive arterial disease of limbs -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary end point of the study was serum creatinine less than 1.5 mg | 15 days

SECONDARY OUTCOMES:
Secondary end points include death of patients | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Singh, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research Chandigarh, Chandigarh, Chandigarh, India

REFERENCES:
- [Result] Alessandria C, Ottobrelli A, Debernardi-Venon W, Todros L, Cerenzia MT, Martini S, Balzola F, Morgando A, Rizzetto M, Marzano A. Noradrenalin vs terlipressin in patients with hepatorenal syndrome: a prospective, randomized, unblinded, pilot study. J Hepatol. 2007 Oct;47(4):499-505. doi: 10.1016/j.jhep.2007.04.010. Epub 2007 May 24. PMID 17560680
- [Derived] Ghosh S, Choudhary NS, Sharma AK, Singh B, Kumar P, Agarwal R, Sharma N, Bhalla A, Chawla YK, Singh V. Noradrenaline vs terlipressin in the treatment of type 2 hepatorenal syndrome: a randomized pilot study. Liver Int. 2013 Sep;33(8):1187-93. doi: 10.1111/liv.12179. Epub 2013 Apr 21. PMID 23601499